CLINICAL TRIAL: NCT06862466
Title: Impact Of An Intervention Education Program On The Knowledge, Attitudes, And Practices Of Dietitians Working With Chronic Kidney Disease Patients In Public Hospitals Of Saudi Arabia
Brief Title: Impact of an Intervention Education Program on the Knowledge, Attitudes, and Practices of Dietitians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Shatha Alattar, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPM-PhDSAlattar
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: No Conditions
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial
Who Masked: Participant
Masking Description: Single (Participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education intervention program (Other): The intervention group will have an education intervention program which will cover five lessons including nutrition assessment for CKD, malnutrition, macro- and micronutrients deficiencies in CKD, nutrition intervention and counselling skills. The education program will be delivered through lectures, workshops, brainstorming and case studies using materials such as PowerPoints, videos, cards, posters, booklets and activities. The program will be offered online via Zoom software, and the learners will have the materials to review at home. The program will be provided in close collaboration between the researcher and the hospital's nutrition department.
  Interventions: Other: Education intervention
- No Intervention: Control group (No Intervention): The control group will not have any intervention.

INTERVENTIONS:
Other: Education intervention — Knowledge, Attitude, and Practice Questionnaire (KAPQ) Regarding Renal Nutrition will be used to collect the data at baseline, after the intervention, and three months follow-up, which is adjusted for clustering.
  Arms: Education intervention program

SUMMARY:
This study aims to develop, implement, and evaluate an educational program-based intervention on the knowledge, attitude, and practice toward renal nutrition among dietitians working with chronic kidney disease (CKD) patients in public hospitals in Saudi Arabia. The study hypothesizes that there will be a significant improvement in the knowledge, attitude, and practice of renal nutrition among the dietitians in the intervention group compared to the control group after the implementation of the educational program. The findings will contribute to enhancing the ability of dietitians to provide effective nutritional care and support for CKD patients in Saudi Arabia.

DETAILED DESCRIPTION:
A cluster randomized controlled trial will be conducted to evaluate the effectiveness of the intervention on the level of knowledge, attitude, and practice in renal nutrition competencies among the dietitians. A total of 100 participants (50 participants for each group) will be select using simple random sampling.

The education intervention program will be developed based on the literature review of the guidelines for the nutritional management of CKD by looking into all evidence-based practice guidelines of renal medical nutrition therapy. The education intervention will include five weeks of in-person education sessions. The education intervention program will cover five lessons including nutrition assessment for CKD, malnutrition, macro- and micronutrients deficiencies in CKD, nutrition intervention and counselling skills. The education program will be delivered through lectures, workshops, brainstorming and case studies using materials such as PowerPoints, videos, cards, posters, booklets and activities. The program will be offered online via Zoom software, and the learners will have the materials to review at home. The program will be provided in close collaboration between the researcher and the hospital's nutrition department.

Data will be collected from four selected public hospitals in Jazan city, Saudi Arabia, by direct interview of the dietitians in the hospitals to determine the competency assessment on knowledge, attitude, and practice of renal nutrition. All respondents in the hospitals will be evaluated before the start of the program (baseline evaluation), after the final intervention session (post-intervention evaluation), and three months after intervention (three-month follow-up after intervention). Data will be analyzed by using the software Statistical Package for Social Sciences (SPSS) version 26.

ELIGIBILITY:
Inclusion Criteria:

* Dietitians who worked with chronic kidney disease patients.
* Dietitians who registered in Saudi Commission for Health Specialties.
* Completed at least one-year experience in their job.
* Dietitians who agree to participate in the study.
* Dietitians who are available at the time of data collection.

Exclusion Criteria:

* Medical doctor dietitians.
* Internship and student.
* Dietitians under one-year experience.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Improved in Knowledge Regarding Renal Nutrition | Timepoint 1 = Baseline. Timepoint 2 = After the intervention (one week post intervention). Timepoint 3 = three months follow-up ( 12 weeks)
  A structured assessment designed to evaluate knowledge and perception of nutrition care including dietary guidelines, nutrient functions, and health benefits will be explored. The assessment consists of 25 questions, each aimed at gauging the respondents' understanding of various aspects of nutrition. Each question will have multiple-choice answers, with one correct answer and several distractors. The best answer will be coded as "1" and the wrong answer as "0". There will be a maximum score of 25 and a minimum of 0.
Improved in Attitude Regarding Renal Nutrition | Timepoint 1 = Baseline. Timepoint 2 = After the intervention (one week post intervention). Timepoint 3 = three months follow-up ( 12 weeks)
  The assessment of attitudes regarding renal nutrition among dietitians will be conducted using a structured questionnaire based on a Likert scale. This approach allows for the quantification of attitudes related to renal diets, which is crucial for evaluating dietitians' perspectives and enhancing their counselling strategies. The proposed questionnaire will consist of 45 questions categorized into five Likert scale options: 1= Never, 2= Rarely, 3=Sometimes, 4 = Often, 5= Always. The scoring system for the questionnaire will range from a minimum score of 45 (if all responses are "Never") to a maximum score of 225 (if all responses are "Always").
Improved in Practice Regarding Renal Nutrition | Timepoint 1 = Baseline. Timepoint 2 = After the intervention (one week post intervention). Timepoint 3 = three months follow-up ( 12 weeks)
  This section involvoes 45 questions related to nutrition care practices. Each question has five possible answers: Never, Rarely, Sometimes, Often, and Always. The response options: Never (1 point), Rarely (2 points), Sometimes (3 points), Often (4 points) and Always (5 points). The total score can range from a minimum of 45 (if all responses are "Never") to a maximum of 225 (if all responses are "Always").

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No